CLINICAL TRIAL: NCT04383782
Title: Examining Outcome Expectancies and Behavioral Reinforcers Among Young Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Responsible Party: Principal Investigator, Amanda Kaufmann, Doctoral Candidate in Clinical Psychology, American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KDYAS2020
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; motivation; outcome expectancies; behavioral reinforcers
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expectancy Challenge (Active Comparator): The expectancy challenge intervention will involve two brief videotaped testimonials in which former smokers discuss their experiences with smoking-related health conditions. Participants will be encouraged to reflect back on the content of each video once per week leading up to the follow-up assessment.
  Interventions: Behavioral: Expectancy Challenge
- Expectancy Challenge + Behavioral Activation (Experimental): In addition to the expectancy challenge intervention (see Expectancy Challenge condition), participants in the Expectancy Challenge + Behavioral Activation group will also receive a novel behavioral activation intervention. Participants will be presented with brief psychoeducation about behavioral activation, several examples of possible functions of cigarette smoking, and several suggestions of behavioral strategies. All participants will receive the same information, but they will be encouraged to apply the information to their personal circumstances and to consider additional examples of rewarding activities they may engage in over the next four weeks. Participants will also be encouraged to engage in at least one behavioral activation activity each week leading up to the follow-up assessment.
  Interventions: Behavioral: Expectancy Challenge + Behavioral Activation
- Neutral Reading (Placebo Comparator): The control group will receive neutral reading materials related to the components and structure of a cigarette. The content will be strictly curated so as to avoid inadvertently encouraging or discouraging smoking among participants.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Expectancy Challenge — Expectancy challenge intervention (see description in study arms).
  Arms: Expectancy Challenge
Behavioral: Expectancy Challenge + Behavioral Activation — Expectancy challenge + behavioral activation interventions (see description in study arms)
  Arms: Expectancy Challenge + Behavioral Activation
Behavioral: Control — Neutral reading condition (see description in study arms).
  Arms: Neutral Reading

SUMMARY:
Chronic cigarette smoking habits often begin in adolescence or early adulthood. 98% of cigarette smokers try their first cigarette before the age of 26. Thus, young adult smokers represent an important target for early smoking cessation intervention. This study tests two interventions designed to increase motivation to quit and decrease smoking behavior. These interventions include: an expectancy challenge approach, which aims to increase negative beliefs about the consequences of smoking; and a behavioral economics approach, which encourages participants to substitute non-smoking behaviors that may still provide reinforcement similar to reinforcement derived from smoking a cigarette.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* English fluency
* Living in the United States
* Smoked at least 1 cigarette per week during the past month
* Willing to be contacted for 1-month follow up assessment

Exclusion Criteria:

* N/A

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
Quit attempt | 4-week follow up
  yes/no, whether or not the participant made a 24-hour (or longer) quit attempt between the date of the main experiment and the date of the 4-week follow-up assessment.
Motivation to quit | 4-week follow up
  Contemplation ladder score (range 0-10; higher scores indicate more motivation to quit)

SECONDARY OUTCOMES:
Smoking rate | 4-week follow up
  past month average self-reported smoking rate
Outcome expectancies | 4-week follow up
  Smoking Consequences Questionnaire (S-SCQ); expected positive and negative consequences of cigarette smoking (range 0-9; higher scores indicate greater positive or negative expectancies)
Behavioral reinforcers | 4-week follow up
  Pleasant Events Schedule (PES); reported behaviors that are pleasurable and not associated with smoking/urge to smoke

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States